CLINICAL TRIAL: NCT04316819
Title: Evaluation of Demonstrations to End Childhood Hunger - CN Food Security
Brief Title: Evaluation of Demonstrations to End Childhood Hunger - CN Food Sec
Acronym: EDECHCNFOODSEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Food and Nutrition Service (U.S. Federal Agency)
Collaborators: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG-3198-C-14-0019 (CN FoodSec)
Record Dates: First submitted 2019-12-12; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Food Insecurity Among Children
Keywords: Food security; Hunger; School children; Indian Tribal Organization; Home-delivered food box

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Packed Promise Demonstration Benefits (Experimental): Treatment households (n=2,143) received one food box per eligible child, per month, delivered to the household, which contained (1) shelf-stable foods, including 6 protein-rich items, 2 dairy items, 4 grain foods, 4 cans of fruit, and 12 cans of vegetables; (2) a nutrition education handout (e.g., a recipe); and (3) a $15 Fresh Check for frozen or fresh fruits and vegetables that participants could redeem at any of 38 Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)-authorized stores or farmers' markets in the study counties.
  Interventions: Other: Packed Promise Demonstration Benefits
- Control Group (No Intervention): Control households (n=2,607) did not receive the treatment benefits but still could participate in other available nutrition assistance programs.

INTERVENTIONS:
Other: Packed Promise Demonstration Benefits — Monthly: Home-delivered food box, nutrition education handout, and $15 monthly voucher for fruits and vegetables
  Arms: Packed Promise Demonstration Benefits

SUMMARY:
The 2010 Child Nutrition Reauthorization provided funding to test innovative strategies to end childhood hunger and food insecurity. Demonstration projects were funded in Chickasaw Nation, Kentucky, Navajo Nation, Nevada, and Virginia. This study focuses on Chickasaw Nation.

School districts were matched, and then one was randomly assigned to either a treatment (n=20) or control group (n=20). Treatment households received one food box per eligible child, per month, delivered to the household, which contained (1) shelf-stable foods, including 6 protein-rich items, 2 dairy items, 4 grain foods, 4 cans of fruit, and 12 cans of vegetables; (2) a nutrition education handout (e.g., a recipe); and (3) a $15 Fresh Check for frozen or fresh fruits and vegetables that participants could redeem at any of 38 Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)-authorized stores or farmers' markets in the study counties. Control households did not receive the treatment benefits but still could participate in other available nutrition assistance programs.

DETAILED DESCRIPTION:
Objective: To reduce childhood food insecurity and hunger, increase families' consumption of nutritious foods, increase the diversity of foods in the home, and ultimately improve diet quality and well-being among children.

Target Population: 40 school districts (115 schools) in 12 counties within the Chickasaw Nation territory in Oklahoma. Within these districts, households with school-age children (both Native American and non-Native American) who were eligible for free school meals or attended a school that participated in the community eligibility provision were eligible to participate in the project.

Intervention School districts were matched, and then one was randomly assigned to either a treatment (n=20) or control group (n=20). Treatment households received one food box per eligible child, per month, delivered to the household, which contained (1) shelf-stable foods, including 6 protein-rich items, 2 dairy items, 4 grain foods, 4 cans of fruit, and 12 cans of vegetables; (2) a nutrition education handout (e.g., a recipe); and (3) a $15 Fresh Check for frozen or fresh fruits and vegetables that participants could redeem at any of 38 Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)-authorized stores or farmers' markets in the study counties. Control households did not receive the treatment benefits but still could participate in other available nutrition assistance programs.

ELIGIBILITY:
Inclusion Criteria:

* 40 school districts (115 schools) in 12 counties within the Chickasaw Nation territory in Oklahoma.
* Within these districts, households with school-age children (both Native American and non-Native American) who were eligible for free National School Lunch Program meals or attended a school that participated in the community eligibility provision were eligible to participate in the project.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4750 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Food Insecurity among Children | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 2 or more out of the 8 child-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.

SECONDARY OUTCOMES:
Very Low Food Insecurity among Children | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 5 or more out of the 8 child-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Food Insecurity among Adults | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 3 or more out of the 10 adult-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Household Food Insecurity | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 3 or more out of the 18 items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Food expenditures | 30 days
  Total amount of Supplemental Nutrition Assistance Program (SNAP) and out-of-pocket food purchases in dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Burke, PhD, Study Director — USDA Food and Nutrition Service

IPD SHARING:
Plan to Share IPD: Yes
Public-use data files are available by request by contacting Michael Burke (michael.burke@usda.gov) or the Office of Policy Support within the USDA Food and Nutrition Service.

REFERENCES:
- [Derived] Briefel RR, Chojnacki GJ, Gabor V, Forrestal SG, Kleinman R, Cabili C, Gleason PM. A Cluster Randomized Controlled Trial of a Home-Delivered Food Box on Food Security in Chickasaw Nation. J Acad Nutr Diet. 2021 Jan;121(1S):S46-S58. doi: 10.1016/j.jand.2020.07.021. PMID 33342524
- See also: Final Report — https://www.fns.usda.gov/ops/evaluation-demonstration-projects-ech